CLINICAL TRIAL: NCT04287101
Title: Home-Based Integrated Post-Acute Care Program for Hip Fracture
Brief Title: Post-acute Care for Patients With Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Shih-Liang Shih, Director of Orthopedics, Taipei City Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAC for hip fracture
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Hip Fractures; Activities of Daily Living
Keywords: Hip fractures; Post-acute care; Home-based care; Hospital-based care; Activities of daily living; Cost effectiveness analysis
MeSH Terms: conditions — Hip Fractures | interventions — Postoperative Period

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- home PAC (Experimental): A home PAC team will care for patients in his/her home within 3 weeks after acute hospitalization. The patient will get a physical therapy (PT) or occupational therapy (OT) 1 to 6 session(s) per week.
  Interventions: Other: Post-operative PT and OT
- hospital PAC (Active Comparator): A rehabilitation PAC team will care for patients in the hospital within 3 weeks after acute hospitalization. The patient will have 1 to 2 session(s) of PT or OT on weekdays, and a daily physician visit and nurse care.
  Interventions: Other: Post-operative PT and OT
- conventional care group (No Intervention): usual care

INTERVENTIONS:
Other: Post-operative PT and OT — Strengthening exercise, range-of-motion exercise, functional training, balance training, adjustment for assistive devices, adaptation and modiﬁcation of the home environment, and patient/caregiver education
  Arms: home PAC; hospital PAC

SUMMARY:
Background and purpose: Hip fracture, a common injury occurred in people aged over 50, may result in disability, poor quality of life, and higher care stress for their families. Aging population and growing number of hip fractures have increased medical expenses, so developed countries implemented post-acute care (PAC) to reduce acute hospitalization, and to improve the quality of care. PAC services can be delivered by hospital/facility-based and home-based services. Previous studies showed that both services could significantly improve patients' activities of daily living and quality of life, and reduce readmissions, long-term care and costs. Taiwan has implemented PAC plan for hip fractures since 2017, but relevant evidences are limited. Therefore, the purpose of this study is to analyze the efficacy and cost-effectiveness of PAC for patients with hip fractures.

DETAILED DESCRIPTION:
Methods: This is a prospective cohort study which will recruit patients aged over 50 with hip fractures receiving surgical treatment in the Taipei City Hospital. They will be provided home-based PAC, hospital-based PAC, or no formal PAC based on the medical judgment and patients/families' willingness. The period of PAC will be two to three weeks after the acute hospitalization. Assessments include physical function (30 seconds sit to stand, Barthel index, and Harris Hip Score), numerical pain rating scale, EuroQol instrument (EQ-5D), Caregiver Strain Index, and using of medical resources. The assessments will be on the day before discharge from acute hospitalization, and on the discharge day from post-acute care. The follow-up assessment will be at 1, 3, 6, and 12 months after operation. The cost-effectiveness ratio will be defined as the New Taiwan dollars paid for 1-unit improvement of functional performance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 50
2. First hip fracture
3. Stable medical condition

Exclusion Criteria:

1. Hip fracture caused by major trauma or pathological condition
2. Multiple fractures
3. Severe physical disability before the hip fracture
4. Unable to cooperate with treatment
5. Further inpatient treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
30-second sit to stand | within 1 year
  Ask participants to cross their arms at the chest, and to perform sit to stand as more as possible within 30 seconds. Measure the repetitions the participants do. Higher repetition indicates more strength of lower extremities.
Activities of daily living Using the Barthel Index (BI) | within 1 year
  Using the Barthel Index (BI) to measure participants' activities of daily living. The self-care domain is self-report by the patient or their families. The mobility domain is observed by the assessor. The greater score indicates more independence.
Functional performance of hip Using the Harris hip score (HHS) | within 1 year
  Using the Harris hip score (HHS) to measure participants' functional performance of hip. The pain domain is self-report by the patient. The function, deformity, and range of motion domain are observed by the assessor. The greater score indicates the better functional performance of hip.
Pain intensity Using the numerical pain rating scale (NPRS) | within 1 year
  Using the numerical pain rating scale (NPRS) to measure participants' pain intensity. Ask participants to report their pain intensity with the 11-point scale (from 0 no pain to 10 worst possible pain).
Quality of lives Using the EuroQol instrument (EQ-5D) | within 1 year
  Part 1: Ask participants to measure their mobility, self-care, usual activities, pain/discomfort, and anxiety/depression with the 3-point scale. The greater score indicates poor quality of life.
Quality of lives Using the EuroQol instrument (EQ-5D) | within 1 year
  Part 2: Ask participants to measure their quality of life with a 20-cm visual analog scale. The greater score indicates a better quality of life.
Caregiver strain Using the caregiver strain index (CSI) | within 1 year
  Using the caregiver strain index (CSI) to measure the strain of caregiver. Ask them to fill a 13-item questionnaire. Greater value indicates a higher strain.
Medical Costs | within 1 year
  Ask participants to record their direct medical cost and indirect medical cost within one year after hip fracture.

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Liang Shih, PhD., Principal Investigator — Department of Orthopaedic, Taipei City Hospital, Zhongxing Branch
Locations (1):
- Taipei City Hospital, Taipei, Taiwan